CLINICAL TRIAL: NCT01083771
Title: Eight Week Plant-based Mediterranean Diet as Prevention of Metabolic Syndrome in Men Undergoing Androgen Deprivation Therapy for Prostate Cancer: A BrUOG Pilot Study
Brief Title: Med Diet Prevention Metabolic Syndrome Men Undergoing Androgen Deprivation Therapy Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BrUOG-MED/PROS-219
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Olive Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olive Oil (Experimental): At least 3 tablespoons of olive oil each day
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Olive Oil — Minimum of 3 tablespoon of olive oil per day

SUMMARY:
The purpose of this study is to assess for changes in a patient's overall energy level and well-being (quality of life) after 8 weeks of dietary intervention.

DETAILED DESCRIPTION:
Primary Objective: To assess for changes in the following measurements after 8 weeks of following a Mediterranean diet-- LDL, HDL, TG, FBS, creatinine, serum testosterone, triglycerides, serum insulin, CRP, 1bs, Waist circumference, blood pressure, body weight

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented carcinoma of the prostate
* On treatment with androgen deprivation therapy for at least 3 months
* Required laboratory values:
* Serum creatinine less than 2.5
* Triglycerides <300
* Fasting glucose < 126
* Testosterone level <50

Exclusion Criteria:

* No diabetes mellitus (Type 1 or 2)
* No renal failure (Serum creatinine > 2.5)
* No active cardiac disease -no history of myocardial infarction/stroke within the last 12 months, no recurrent unstable angina, uncontrolled/unstable arrhythmias, uncontrolled hypertension (systolic blood pressure >160, diastolic blood pressure >100)
* No severe peripheral vascular disease
* No commencement of lipid lowering agent within 8 weeks of enrollment the study or change in dose throughout the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mega, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olive Oil
Started | 21
Completed | 16
Not Completed | 5
Not completed — non-compliant | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Olive Oil
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 69.9 [58 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Blood Chemistry (Fasting Triglycerides) After 8 Weeks of Following a Mediterranean Diet
Description: Based on overall percentage change at baseline versus post diet
Time Frame: eight weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Olive Oil
Number analyzed (Participants) | 21
percentage of change | 21 (38.2)

2. Secondary Outcome: To Assess Changes in the Body After 8 Weeks of Following a Mediterranean Diet
Description: Post diet waist circumference
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Olive Oil
Number analyzed (Participants) | 21
centimeters | 102.4 (8.8)

ADVERSE EVENTS:
Arm/Group | Olive Oil
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olive Oil (N=21)
Chest pain (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olive Oil (N=21)
creatinine increased (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No